CLINICAL TRIAL: NCT05172687
Title: The Effect of De-Prescribing Antipsychotics on Health and Quality of Life for People With Dementia
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Bureau of Economic Research, Inc. (Other); Harvard School of Public Health (HSPH) (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Adam Sacarny, PhD, Assistant Professor of Health Policy and Management, Columbia University
Other Study IDs: AAAT2250; R21AG070942 (NIH)
Record Dates: First submitted 2021-12-13; First posted 2021-12-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease; Dementia; Prescribing, Off-Label
Keywords: antipsychotics; alzheimers; dementia; prescribing; deprescribing; nursing homes; long-term care
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Nursing home patients of treated study prescribers: Patients attributed to physicians who received overprescribing letters in the primary study who reside in a nursing home.
  Interventions: Behavioral: Overprescribing letter to attributed physician
- Nursing home patients of control study prescribers: Patients attributed to physicians who received placebo letters in the primary study who reside in a nursing home.
  Interventions: Behavioral: Placebo letter to attributed physician
- Community-dwelling patients of treated study prescribers: Patients attributed to physicians who received overprescribing letters in the primary study who reside in the community.
  Interventions: Behavioral: Overprescribing letter to attributed physician
- Community-dwelling patients of control study prescribers: Patients attributed to physicians who received placebo letters in the primary study who reside in the community.
  Interventions: Behavioral: Placebo letter to attributed physician

INTERVENTIONS:
Behavioral: Overprescribing letter to attributed physician — Letter telling patient's attributed physician they were under review for high prescribing
  Groups: Community-dwelling patients of treated study prescribers; Nursing home patients of treated study prescribers
Behavioral: Placebo letter to attributed physician — Letter to patient's attributed physician about unrelated Medicare regulation
  Groups: Community-dwelling patients of control study prescribers; Nursing home patients of control study prescribers

SUMMARY:
This study aims to analyze how warning letters sent to physicians prescribing high levels of the antipsychotic quetiapine affected the health and quality of life of their patients with dementia. Using a randomized controlled trial conducted by the Centers for Medicare and Medicaid Services (CMS) in 2015, this secondary study looks at the effects of potential de-prescribing of antipsychotics by study physicians induced by the letters. The central question is whether the intervention led to better health and quality of life outcomes by encouraging more guideline-concordant care and whether changes in physicians' prescription behavior caused unintended harms.

ELIGIBILITY:
Inclusion Criteria:

* Fully enrolled in Fee-For-Service Medicare Parts A, B, and D
* For nursing home patients: Residing in a nursing home and has a usable nursing home assessment to measure outcomes
* For community-dwelling patients: Not residing in a nursing home
* Has Alzheimer's or dementia related disease diagnosis
* Attributed to study physician (see study population description)

Exclusion Criteria:

* Died during 90 day period used to attribute patient to physician
* For nursing home patients: Short-stay nursing facility patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Repeated cross sections of patients attributed to study prescribers. Analyses are conducted separately for patients residing in nursing homes and patients living in the community. The investigators look at a series of sequential 90 day periods with the first period beginning at the start of the intervention. The investigators measure outcomes based on health care assessments, encounters, and claims that occur during the period. The investigators attribute patients to study prescribers based on their evaluation and management encounters during the 90 days preceding the period for nursing home patients and during the 180 days preceding the period for community-dwelling patients. The patient is attributed to the physician who rendered the most of these services.
Sampling Method: Non-Probability Sample
Enrollment: 336460 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Days of Quetiapine Received | 90 days
  Days of quetiapine received during the outcome measurement period

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sacarny, PhD, Principal Investigator — Columbia University; Michael L Barnett, MD, MS, Study Director — Harvard School of Public Health (HSPH)
Locations (3):
- United States (3):
  - Harvard T.H. Chan School of Public Health, Boston, Massachusetts
  - National Bureau of Economic Research, Cambridge, Massachusetts
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No
Because this study uses restricted-access Medicare data, we will not be able to share individual participant data.

REFERENCES:
- [Derived] Harnisch M, Barnett ML, Coussens S, Thomas KS, Olfson M, Berhane K, Sacarny A. Physician Antipsychotic Overprescribing Letters and Cognitive, Behavioral, and Physical Health Outcomes Among People With Dementia: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e247604. doi: 10.1001/jamanetworkopen.2024.7604. PMID 38662373
- See also: ClinicalTrials.gov entry for original randomized trial — https://clinicaltrials.gov/ct2/show/NCT02467933
- See also: OSF.io Project Page — https://osf.io/eh47k/